CLINICAL TRIAL: NCT04879875
Title: New Method for Real-time Detection of Tissue Ischemia; IscAlert™ - Study
Brief Title: New Method for Real-time Detection of Tissue Ischemia (ISCALERT)
Acronym: ISCALERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Magne Røkkum, Head Orthopaedic Department/Professor, Oslo University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-21
Record Dates: First submitted 2021-04-27; First posted 2021-05-10 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Ischemia; Blood Circulation Disorder; Carbon Dioxide; Biosensing Techniques
Keywords: Ischemia; Carbon dioxide; Biosensor; Musculature; Subcutaneous; Surgery; Orthopedic; Limb
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Intervention Model Description: Prospective, Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients scheduled for limb (arm/leg) surgery with tourniquet where IscAlert is removed immediately after surgery.
  All patients will receive 3 sensors in the limb undergoing surgery and two control sensors in the opposite limb. The sensor in the opposite extremity which is not to be operated serves as a reference value for CO2.
  Interventions: Device: IscAlert
- Group 2 (Experimental): Patients scheduled for limb (arm/leg) surgery with tourniquet where IscAlert is removed 72 hours after surgery.
  All patients will receive 3 sensors in the limb undergoing surgery and two control sensors in the opposite limb. The sensor in the opposite extremity which is not to be operated serves as a reference value for CO2.
  Interventions: Device: IscAlert 72h

INTERVENTIONS:
Device: IscAlert — 3 IscAlert sensors in the limb undergoing surgery and two control sensors in the opposite limb are inserted and CO2 is measured continously. IscAlert sensors are removed after end of surgery.
  Arms: Group 1
Device: IscAlert 72h — 3 IscAlert sensors in the limb undergoing surgery and two control sensors in the opposite limb are inserted and CO2 is measured continously. IscAlert sensors are removed 72 hours after end of surgery
  Arms: Group 2

SUMMARY:
This is a prospective, single arm, open, single centre clinical investigation designed to examine the feasibility and safety of the IscAlert™ device in patients scheduled for limb (arm/leg) surgery with tourniquet. IscAlert is measuring CO2 in muscular and subcutaneous tissue. IscAlert is inserted into normal muscle and subcutaneous tissue in ischemic (operated limb with a tourniquet) and non-ischemic limb (non-operated limb).After the tourniquet is inflated, ischemia develops in the muscles and subcutaneous tissue. This will result in an increase in CO2, which will be detected by the sensors on the operated extremity, while the sensors on the non-operated will show normal values. After releasing the tourniquet cuff, the muscle will be reperfused and the CO2 level is expected to decrease into normal levels. 50 number of patients will be enrolled to undergo the procedures. The IscAlert will be removed from the patient before the patient is discharged from the operating room, but in 25 of the patients, IscAlert™ will be inserted for 72 hours in the operated extremity after the end of surgery. After this, the sensors are removed. 250 Devices is planned to be used in this clinical study.

DETAILED DESCRIPTION:
This is a prospective, single arm, open, single centre clinical investigation designed to examine the feasibility and safety of the IscAlert™ device in patients scheduled for limb (arm/leg) surgery with tourniquet.

50 number of patients will be enrolled to undergo the procedures detailed in this clinical investigational plan using 250 devices.

IscAlert is 0.8 mm in diameter and in vitro testing, shows stable and accurate measurements of pCO2. More than 100 animal experiments have been done with the sensor. The experiments have shown that the sensor detects ischemia (Increased CO2-measurements) in real time in the following organs and tissues: Brain, heart, liver, kidneys, pancreas, intestines, musculature and subcutaneous tissue. Sensitivity and specificity are close to 100%. The sensors are inserted into tissue by a split needle technique. The split needle is the size of a 3-gauge peripheral venous catheter. In animal studies, no complications have been detected when using the sensor.

The IscAlert catheters are connected to an electronics unit that is fixed to the skin with an adhesive plaster outside the sterile area. The electrical signals are redirected to a PC approved for clinical use which continuously records tissue pressures of CO2.

IscAlert sensors (3 - three) are inserted into normal muscle and subcutaneous tissue proximal on the limb to be operated. The insertion is distal to the blood cuff, and far away from the surgery field. The insertion is done under sterile conditions in accordance with standard sterility criteria at the hospital. No pain during insertion will occur because of insertion is performed after anesthesia induction. Also, the insertion can be compared to an intramuscular injection.

Two identical IscAlert sensors are also inserted in the opposite extremity that is not to be operated and serves as a reference value. After the tourniquet is inflated, ischemia develops in the muscles and subcutaneous tissue. This will result in an increase in CO2, which will be detected by the sensors on the operated extremity, while the sensors on the non-operated will show normal values.

After releasing the tourniquet cuff, the muscle will be reperfused and the CO2 level is expected to decrease into normal levels within 15 - 45 minutes. In 25 patients, the biosensors will be removed from the patient before the patient is discharged from the operating room, but in 25 of the patients, IscAlert will be inserted for up to 72 hours in the operated extremity after the end of surgery to identify drifting of the sensors. After this, the sensors are removed.

The primary objective is to evaluate the ability of the IscAlert device to measure CO2-levels in ischemic and non-ischemic limb musculature and subcutaneous tissue in patients who experience orthopedic surgery with limb tourniquet and to assess the safety/efficacy using device IscAlert.

Our hypotheses are:

The IscAlert device will be able to detect the presence of ischemia in muscle and subcutaneous tissue, whereby CO2 levels, measured by IscAlert, will be higher in ischemic musculature than non-ischemic musculature in patients undergoing orthopedic limb surgery.

No clinically significant bleeding or infection will occur using IscAlert in this clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be scheduled for orthopedic limb surgery with planned use of tourniquet.
* Subject must be ≥ 18 years
* Able to give written signed informed consent
* Tourniquet planned to be used > 30 minutes

Exclusion Criteria:

* Sign of inflammation/infection, hematoma, and traumatized tissue at insertion site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-07-24 (Actual)

PRIMARY OUTCOMES:
Tissue CO2-level | 72 hours
  Tissue CO2-level (kPa) during insertion periode

SECONDARY OUTCOMES:
Bleeding | 72 hours
  Amount of blood from insertion site (ml)
Infection | 30 days
  Infection from insertion site at the discretion of the investigator (yes or no)
Pain score at insertion site - Numerical Rating Scale (NRS) - 30 days after discharge from hospital | 30 days
  Pain from insertion site measured by Numeric Rating Scale (NRS; 0-10 points)
Pain score at insertion site - Numerical Rating Scale (NRS) - 7 days after discharge from hospital | 7 days
  Pain from insertion site measured by Numeric Rating Scale (NRS; 0-10 points)
Arterial CO2 level | 3 hours
  Blood gass analysis of CO2 during surgery (kPa)
Arterial lactate level | 3 hours
  Blood gass analysis of lactate during surgery (mmol/L)
Arterial pH level | 3 hours
  Blood gass analysis of pH during surgery
Arterial O2 level | 3 hours
  Blood gass analysis of O2 during surgery (Kpa)
Time of tourniquet | 180 minutes
  Minutes of inflated tourniquet during surgery (minutes)
End-tidal level of CO2 | 4 hours
  End-tidal level of CO2 during anesthesia (kPa)
End-tidal level of CO2 72 hours | 72 hours
  End-tidal level of CO2 during postoperative recovery (kPa)
Duration of surgery | 180 minutes
  Duration of surgery - Number of minutes
Duration of anesthesia | 240 minutes
  Duration of anesthesia - Number of minutes

CONTACTS AND LOCATIONS:
Overall Officials: Magne Røkkum, Ph.d., Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD to other researchers